CLINICAL TRIAL: NCT05604638
Title: Safety and Efficacy of Early Administration of Tirofiban in Patients Treated With Tenecteplase for Acute Ischemic Stroke
Brief Title: Early Administration of Tirofiban in Patients Treated With Tenecteplase for Acute Ischemic Stroke
Acronym: INSTANT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: Ganzhou People's Hospital (Unknown)
Responsible Party: Principal Investigator, Jian Zhang, MD, Research assistant, Second Affiliated Hospital of Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SecondAHGuangxiMU
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
Keywords: randomized trial; tenecteplase; tirofiban; intravenous thrombolysis
MeSH Terms: conditions — Ischemic Stroke | interventions — Tirofiban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban (Experimental): Patients are treated with intravenous tenecteplase first, and patients who meet the selection criteria will be randomly assigned to either the tirofiban or placebo group in a 1:1 ratio. Patients assigned to the tirofiban group will be treated with intravenous tirofiban. It is recommended to start treatment as soon as possible (within 10 minutes recommended) after randomization. Tirofiban will be administered at a dose of 0.3 μg per kilogram of body weight per minute for 30 minutes, followed by a continuous infusion of 0.075 μg per kilogram per minute for 47.5h. Aspirin placebo (1 tablet) and/or clopidogrel placebo (1 tablet) will be given orally at 24h after intravenous tenecteplase. Antiplatelet therapy with aspirin (100 mg) and/or clopidogrel (75 mg) will be administered at 44h after randomization until the follow-up period of 90 days.
  Interventions: Drug: Tirofiban Hydrochloride
- Placebo (Placebo Comparator): All patients are treated with intravenous tenecteplase first, and patients who meet the selection criteria will be randomly assigned to either the tirofiban or placebo group in a 1:1 ratio. Patients assigned to the placebo group will be treated with intravenous saline. It is recommended to start treatment as soon as possible (within 10 minutes recommended) after randomization. Placebo will be administered at a dose of 0.3 μg per kilogram of body weight per minute for 30 minutes, followed by a continuous infusion of 0.075 μg per kilogram per minute for 47.5h. Aspirin (1 tablet) and/or clopidogrel (1 tablet) will be given orally at 24h after intravenous tenecteplase. Antiplatelet therapy with aspirin (100 mg) and/or clopidogrel (75 mg) will be administered at 44h after randomization until the follow-up period of 90 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirofiban Hydrochloride — Patients will receive a continuous intravenous infusion of tirofiban at a dose of 0.3 μg per kilogram of body weight per minute for 30 minutes, followed by a continuous infusion of 0.075 μg per kilogram per minute for 47.5h after start of tenecteplase treatment within 4-24 hours. Aspirin placebo (1 tablet) and/or clopidogrel placebo (1 tablet) will be given orally at 24h after intravenous tenecteplase. Antiplatelet therapy with aspirin (100 mg) and/or clopidogrel (75 mg) will be administered at 44h after randomization until the follow-up period of 90 days.
  Arms: Tirofiban
Drug: Placebo — Patients will receive a continuous intravenous infusion of placebo at a dose of 0.3 μg per kilogram of body weight per minute for 30 minutes, followed by a continuous infusion of 0.075 μg per kilogram per minute for 47.5h after start of tenecteplase treatment within 4-24 hours. Aspirin (1 tablet) and/or clopidogrel (1 tablet) will be given orally at 24h after intravenous tenecteplase. Antiplatelet therapy with aspirin (100 mg) and/or clopidogrel (75 mg) will be administered at 44h after randomization until the follow-up period of 90 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of early administration of tirofiban in patients treated with tenecteplase for acute ischemic stroke.

DETAILED DESCRIPTION:
Intravenous thrombolysis with alteplase is recommended in treatment guidelines for patients with acute ischemic stroke. Previous studies showed that intravenous tenecteplase (0.25 mg/kg) is a reasonable alternative to alteplase for all patients presenting with acute ischemic stroke who meet standard criteria for thrombolysis. After thrombolysis-induced recanalisation, reocclusion occurs in 14-34% of patients, probably because of platelet activation. Early administration of antiplatelet therapy after intravenous thrombolysis could reduce the risk of reocclusion and improve outcome. The purpose of this study is to assess the safety and efficacy of early administration of tirofiban in patients treated with tenecteplase for acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Within 4-24 hours after intravenous thrombolytic therapy with tenerplase for acute ischemic stroke, there was no significant change in symptoms compared to the baseline (defined as an increase or decrease of 0 or 1 point in the NIHSS score), and neurological function deteriorated (defined as an increase of ≥ 2 in the NIHSS score compared to the baseline) Fluctuations in neurological function (defined as an increase of 4 points or more in the NIHSS score compared to the baseline and then a decrease of 4 points or more);
3. NIHSS ≥ 4 points before randomization;
4. The patient or their family members sign a written informed consent form.

Exclusion Criteria:

1. Intracranial hemorrhage was confirmed by CT or MRI after intravenous thrombolysis and before randomization;
2. CTA/MRA/DSA showed occlusion of the internal carotid artery, middle cerebral artery M1, M2 or M3 segment, anterior cerebral artery A1, A2 or A3 segment, posterior cerebral artery P1, P2 or P3, vertebral or basilar artery;
3. Confirmed or suspected cardioembolic stroke mechanisms, including any of the following: documented cardiac sources of thromboembolism: chronic or paroxysmal atrial fibrillation, rheumatic mitral stenosis, prosthetic heart valves, infective endocarditis, intracardiac thrombus or implanted prosthetic material, dilated cardiomyopathy (left ventricular ejection fraction <40%), or spontaneous echo contrast in the left atrium; other laboratory-confirmed embolic sources: patent foramen ovale with concomitant atrial septal aneurysm, or cryptogenic stroke with a CHADS-VASC score ≥ 2 indicating high thromboembolic risk;
4. Blood platelet count was lower than 100×10^9/L;
5. Renal insufficiency, glomerular filtration rate < 30 mL/min;
6. Pregnant or lactating women;
7. Allergic to tirofiban, nickel, titanium or their alloys;
8. Prior neurological or psychiatric illness that prevents assessment of neurological function;
9. Pre-existing bleeding disease, severe heart, liver, or kidney disease, or sepsis;
10. Brain tumors with a space-occupying effect on imaging (other than micromeningiomas);
11. Intracranial aneurysm, arteriovenous malformation;
12. Life expectancy of any advanced disease < 6 months;
13. Participating in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Excellent functional outcome | 90 days post-randomization
  modified Rankin scale score of 0 to 1. modified Rankin scale scores range from 0 to 6, with 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death.

SECONDARY OUTCOMES:
Ordinal degree of disability | 90 days post-randomization
  Ordinal degree of disability on the modified Rankin scale score at 90 days (shift analysis)
Functionally independent | 90 days post-randomization
  modified Rankin scale score of 0 to 2
Ambulatory or bodily needs capable or better | 90 days post-randomization
  modified Rankin scale score of 0 to 3
Early neurologic improvement | 48 hours post-randomization
  defined as the National Institutes of Health Stroke Scale score at 48 hours after randomization, is reduced by 30% or more compared to the National Institutes of Health Stroke Scale score at randomization
Health-related quality of life | 90 days post-randomization
  assessed with the European Quality Five Dimensions Five Level scale
Symptomatic intracranial hemorrhage | 48 hours post-randomization
  defined as per the Heidelberg bleeding classification
Radiologic intracranial hemorrhage rate | 48 hours post-randomization
  diagnosed with intracranial hemorrhage (including bleeding in brain parenchyma, subarachnoid space, etc.) via radiologic examinations (e.g., computed tomography or magnetic resonance imaging
Mortality | 90 days post-randomization
  The proportion of participants who die from any cause within 90 days after randomization in the study
Incidence of non-hemorrhagic serious adverse events | Within 90 days post-randomization
  such as pneumonia, respiratory failure, circulatory failure, cerebral herniation, secondary epilepsy, sepsis, renal failure, acute coronary syndrome, venous thrombosis, etc
Other serious adverse events | Within 90 days post-randomization
  Serious adverse events that are not categorized as non-hemorrhagic (as listed in Outcome 10), including any unlisted severe medical events requiring medical intervention or leading to significant clinical deterioration

OTHER OUTCOMES:
Ordinal degree of disability | 1 year post-randomization
  Ordinal degree of disability on the modified Rankin scale score at 1 year (shift analysis)
Excellent functional status | 1 year post-randomization
  modified Rankin scale score 0 to 1 at 1 year
Functionally independent | 1 year post-randomization
  modified Rankin scale score 0 to 2 at 1 year
Ambulatory or bodily needs capable or better | 1 year post-randomization
  modified Rankin scale score 0 to 3 at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhongming Qiu, MD, Principal Investigator — Sun Yet-sen University
Locations (38):
- China (38):
  - Mingguang People's Hospital, Chuzhou, Anhui
  - Longyan People´s Hospital, Longyan City, Longyan, Fujian
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Huangmei People's Hospital, Huanggang, Hubei
  - Yiling People's Hospital of Yichang city, Yichang, Hubei
  - Hunan Xupu Chengnan Hospital, Huaihua, Hunan
  - People's Hospital Of Shaodong, Shaoyang, Hunan
  - Shaoshan People's Hospital, Xiangtan, Hunan
  - Xiangtan Central Hospitall, Xiangtan, Hunan
  - Hunan University of Medicine Affiliated Pingjiang Hospital, Yueyang, Hunan
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - People's Hospital of Dayu County, Ganzhou, Jiangxi
  - People's Hospital of Ganxian District, Ganzhou, Jiangxi
  - People's Hospital of Quannan County, Ganzhou, Jiangxi
  - People's Hospital of RuiJin City, Ganzhou, Jiangxi
  - People's Hospital of Shangyou County, Ganzhou, Jiangxi
  - People's Hospital of Xinfeng County, Ganzhou, Jiangxi
  - People's Hospital of Xunwu County, Ganzhou, Jiangxi
  - People's Hospital of Yudu County, Ganzhou, Jiangxi
  - Ganzhou Municipal Hospital, Ganzhou, Jiangxi
  - Nankang TCM Hospital, Ganzhou, Jiangxi
  - People's Hospital of Anyuan County, Ganzhou, Jiangxi
  - People's Hospital of Chongyi County, Ganzhou, Jiangxi
  - People's Hospital of Shicheng County, Ganzhou, Jiangxi
  - Second Hospital of Xingguo County, Ganzhou, Jiangxi
  - Second People's Hospital of Yudu County, Ganzhou, Jiangxi
  - The People's Hospital of Ningdu County, Ganzhou, Jiangxi
  - Traditional Chinese Medicine Hospital of Xingguo County, Ganzhou, Jiangxi
  - Traditional Chinese Medicine Hospital of Yudu County, Ganzhou, Jiangxi
  - Affiliated Hospital of Jiujiang University, Jiujiang, Jiangxi
  - Ji'an Central People's Hospital, Ji’an, Jiangxi
  - People's Hospital of Wan'an county, Ji’an, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - People's Hospital of Yichun, Yichun, Jiangxi
  - Yingtan People's Hospital, Yingtan, Jiangxi
  - Songyuan Jilin Oilfield Hospital, Songyuan, Jilin
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - Zhongmeng Hospital of Hexigten Banner, Chifeng, Neimenggu

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan, and Analytic Code will be shared after approval of a proposal from principal investigator 3 years after the trial results are revealed.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 3 years after the trial results are revealed.
Access Criteria: After approval of a proposal from principal investigator
URL: http://hsyygy@163.com